CLINICAL TRIAL: NCT03538691
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled Trial to Evaluate the Efficacy, Safety, and Tolerability of Brexpiprazole as Adjunctive Therapy in the Maintenance Treatment of Adults With Major Depressive Disorder
Brief Title: A Trial to Evaluate the Efficacy, Safety & Tolerability of Brexpiprazole in the Maintenance Treatment of Adults With Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 331-201-00079; 2018-000601-22 (EudraCT Number)
Record Dates: First submitted 2018-04-13; First posted 2018-05-29 (Actual); Results first posted 2023-10-12 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Major Depressive Disorder
Keywords: Brexpiprazole; MDD
MeSH Terms: conditions — Depressive Disorder, Major | interventions — brexpiprazole

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase A: Brexpiprazole + ADT (Experimental): Participants received brexpiprazole 2 or 3 milligrams per day (mg/day) along with protocol-specified antidepressant therapy (ADT), orally, for 6 to 8 weeks during Phase A. Participants were initially titrated to a target dose of brexpiprazole 2 mg over a 2 to 4-week period. Thereafter, participants who had not met response criteria as defined in the blinded addendum, did not have potentially dose-related adverse events (AEs), and had not achieved the maximum dose of medication had their dose increased up to 3 mg.
  Interventions: Drug: Brexpiprazole; Drug: Antidepressant therapy
- Phase B: Brexpiprazole + ADT (Experimental): Eligible participants completing Phase A were enrolled in Phase B to receive brexpiprazole 2 or 3 mg/day along with protocol-specified ADT, orally, for 12 weeks.
  Interventions: Drug: Brexpiprazole; Drug: Antidepressant therapy
- Phase C: Brexpiprazole + ADT (Experimental): Eligible participants completing Phase B received brexpiprazole 2 or 3 mg/day (dose of brexpiprazole that they were receiving at Week 20 of the Stabilization Phase) along with protocol-specified ADT, orally, for up to 26 weeks during Phase C.
  Interventions: Drug: Brexpiprazole; Drug: Antidepressant therapy
- Phase C: Placebo + ADT (Experimental): Eligible participants completing Phase B received brexpiprazole-matching placebo along with protocol-specified ADT, orally, for up to 26 weeks during Phase C.
  Interventions: Drug: Antidepressant therapy

INTERVENTIONS:
Drug: Brexpiprazole — Administered as tablets.
  Other Names: OPC-34712; Rexulti
  Arms: Phase A: Brexpiprazole + ADT; Phase B: Brexpiprazole + ADT; Phase C: Brexpiprazole + ADT
Drug: Antidepressant therapy — Protocol-specified oral ADTs included:
  citalopram hydrobromide (Celexa®) tablets, escitalopram (Lexapro®) tablets, fluoxetine (Prozac®) capsules, paroxetine (Paxil CR®) controlled-release tablets, sertraline (Zoloft®) tablets, duloxetine (Cymbalta®) delayed-release capsules, venlafaxine XR (Effexor XR®) extended-release (XR) capsules.

SUMMARY:
Major depressive disorder (MDD) is a serious medical illness associated with significant suicidal risk and marked disability. Despite the availability of numerous treatments, achievement of consistent and favorable long-term outcomes remains challenging.

This study will assess the safety, efficacy and tolerability of brexpiprazole as adjunctive therapy to protocol-specific open-label antidepressant therapy.

ELIGIBILITY:
Inclusion Criteria:

* Participants with both a diagnosis of recurrent major depressive disorder, and in a current major depressive episode of ≥ 8 weeks in duration, as defined by Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) and confirmed by both the Mini International Neuropsychiatric Interview (MINI) and an adequate clinical psychiatric evaluation.
* Participants must have reported a history for the current major depressive episode of an inadequate response to 1 or 2 adequate antidepressant treatments, and participants must currently be taking a protocol-mandated antidepressant treatment at an adequate dose and duration, and most not have reported ≥ 50% improvement. For participants who are currently on an adequate dose of protocol-mandated antidepressant therapy (ADT), but for an inadequate duration, can use the screening period to achieve adequate duration. At Phase A baseline visit, all participants must have either 2 or 3 documented inadequate responses to antidepressant treatment in total for the current episode as defined by the Massachusetts General Hospital Antidepressant Treatment Response Questionnaire (ATRQ).
* Participants with a Hamilton Rating Scale for Depression (HAM-D17) total score ≥ 18 at the screening visit, and Phase A baseline visits.
* Participants willing to discontinue all prohibited psychotropic medications to meet protocol-required washouts prior to and during the trial period.

Exclusion Criteria:

* Females who are breast-feeding and/or who have a positive pregnancy test result prior to receiving investigational medicinal product (IMP).
* Sexually active males or females of childbearing potential who do not agree to practice 2 different methods of birth control or remain abstinent during the trial and for 30 days after the last dose of IMP.
* Participants who report treatment with adjunctive antipsychotic medication with an antidepressant for a minimum of 3 weeks during the current major depressive episode.
* Participants who report allergies or an intolerability (lifetime treatment history) to trial-provided ADTs that have not been prescribed to the participant during the current major depressive episode.
* Participants who have received electroconvulsive therapy (ECT) for the current major depressive episode.
* Participants who have had an inadequate response to ECT at any time in the past or who have had a vagus nerve stimulation or deep brain stimulation device implanted at any time for the management of treatment-resistant depression. Participants who have had transcranial magnetic stimulation during the current major depressive episode.
* Participants with a current need for involuntary commitment or who have been hospitalized within 4 weeks of screening for the current major depressive episode.
* Participants with a primary DSM-5 diagnosis of:

  1. Schizophrenia Spectrum and Other Psychotic Disorders
  2. Bipolar and Related Disorders
  3. Obsessive Compulsive Disorders
  4. Feeding and Eating Disorders
  5. Neurocognitive Disorders
  6. Panic Disorder
  7. Post-Traumatic Stress Disorder
* Participants with a current DSM-5 diagnosis of borderline, antisocial, paranoid, schizoid, schizotypal, or histrionic personality disorder or intellectual disability.
* Participants experiencing hallucinations, delusions, or any psychotic symptomatology in the current major depressive episode.
* Participants receiving new onset psychotherapy (individual, group, marriage or family therapy) within 42 days of screening or at any time during participation in the trial.
* Participants who have met DSM-5 criteria for substance use disorder (moderate or severe) within the past 60 days; including alcohol and benzodiazepines, but excluding nicotine.
* Participants with hypothyroidism or hyperthyroidism (unless condition has been stabilized with medications for at least the past 90 days) and/or an abnormal result for free T4 at screening.
* Participants who currently have clinically significant neurological, hepatic, renal, metabolic, hematological, immunological, cardiovascular, pulmonary, or gastrointestinal disorders such as any history of myocardial infarction, congestive heart failure, HIV seropositive status/acquired immunodeficiency syndrome, chronic hepatitis B or C.
* Participants with diabetes mellitus (IDDM and non-IDDM) are ineligible for the trial unless their condition is stable and well-controlled.
* Participants with uncontrolled hypertension (DBP > 95 millimetres of mercury [mmHg]) or symptomatic hypotension, or orthostatic hypotension which is defined as a decrease of ≥ 30 mmHg in systolic blood pressure (SBP) and/or decrease of ≥ 20 mmHg in diastolic blood pressure (DBP) after at least 3 minutes standing compared to the previous supine blood pressure OR development of symptoms.
* Participants with known ischemic heart disease or history of myocardial infarction-or congestive heart failure (whether controlled or uncontrolled).
* Participants with epilepsy or a history of seizures, except for a single seizure episode.
* Participants with a positive drug screen for cocaine or other drugs of abuse (excluding known prescription stimulants and other medications and marijuana). Detectable levels of alcohol, marijuana, barbiturates, or opiates in the drug screen are not exclusionary if, in the investigator's documented opinion, the participant does not meet DSM-5 criteria for moderate to severe substance use disorder and the positive test does not signal a clinical condition that would impact the safety of the participant or interpretation of the trial results, and participation is agreed to by the medical monitor prior to treatment.
* Treatment with a monoamine oxidase inhibitor (MAOI) within 14 day prior to the first dose of IMP in Phase A.
* Use of benzodiazepines and/or hypnotics (including non-benzodiazepine sleep aids) within 7 days prior to first dose of IMP in Phase A.
* Use of varenicline within 5 days prior to the first dose of IMP in Phase A.
* Use of oral (or immediate release intramuscular) neuroleptics within 7 days prior or long-acting approved neuroleptics ≤ 1 full cycle plus 1/2 cycle prior to the first dose of IMP in Phase A.
* Participants who would be likely to require prohibited concomitant therapy during the trial.
* Participants who have been exposed to brexpiprazole in any prior clinical trial or has received commercial brexpiprazole (Rexulti).
* Participants with a history of neuroleptic malignant syndrome or serotonin syndrome.
* Participants with a history of true allergic response to more than one class of medications.
* Prisoners or participants who are compulsorily detained for treatment of either a psychiatric or physical illness.
* Participants who participated in any clinical trial within the last 60 days or who participated in more than 2 clinical trials within the past year.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1149 (Actual)
Dates: Start 2018-07-13 (Actual); Primary Completion 2022-07-08 (Actual); Study Completion 2022-07-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- For additional information regarding sites, contact 844-687-8522, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on the Vivli data sharing platform which can be found here: https://vivli.org/ourmember/Otsuka/
URL: https://clinical-trials.otsuka.com

REFERENCES:
- [Derived] McIntyre RS, Sundararajan K, Behl S, Hefting N, Jin N, Brewer C, Hobart M, Thase ME. A double-blind, placebo-controlled, randomised withdrawal study of adjunctive brexpiprazole maintenance treatment for major depressive disorder. Acta Neuropsychiatr. 2024 Oct 17;37:e33. doi: 10.1017/neu.2024.32. PMID 39415650

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1149 participants with major depressive disorder (MDD) participated in the study from 13 July 2018 to 29 July 2022.
Pre-assignment Details: Of the 1149 participants enrolled in Phase A (Acute Treatment) of the study, 766 eligible participants continued to Phase B (Stabilization). Eligible participants who completed the Phase B were randomized into Phase C (Double-blind Randomized Withdrawal) to receive brexpiprazole or placebo along with open-label antidepressant therapy (ADT) in a 1:1 ratio for up to 26 weeks.
Period: Phase A: Acute Treatment (up to 8 Weeks)
Arm/Group | Phase A: Brexpiprazole + ADT | Phase B: Brexpiprazole + ADT | Phase C: Brexpiprazole + ADT | Phase C: Placebo + ADT
Started | 1149 | 0 | 0 | 0
Phase A Safety Sample (The Phase A Safety Sample included all participants who received at least 1 dose of brexpiprazole in Phase A.) | 1136 | 0 | 0 | 0
Completed | 766 | 0 | 0 | 0
Not Completed | 383 | 0 | 0 | 0
Not completed — Lost to Follow-up | 24 | 0 | 0 | 0
Not completed — Adverse Event | 82 | 0 | 0 | 0
Not completed — Subject Withdrew Consent | 54 | 0 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0
Not completed — Non-Compliance With Study Drug | 9 | 0 | 0 | 0
Not completed — Lack of Efficacy | 185 | 0 | 0 | 0
Not completed — Protocol Deviation | 12 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0
Not completed — Reason not Specified (not due to Coronavirus Disease 2019 [COVID-19] Restriction) | 15 | 0 | 0 | 0
Period: Phase B: Stabilization (12 Weeks)
Arm/Group | Phase A: Brexpiprazole + ADT | Phase B: Brexpiprazole + ADT | Phase C: Brexpiprazole + ADT | Phase C: Placebo + ADT
Started | 0 | 766 | 0 | 0
Phase B Safety Sample (The Phase B Safety Sample included all participants who received at least 1 dose of brexpiprazole in Phase B.) | 0 | 765 | 0 | 0
Completed | 0 | 489 | 0 | 0
Not Completed | 0 | 277 | 0 | 0
Not completed — Lost to Follow-up | 0 | 5 | 0 | 0
Not completed — Adverse Event | 0 | 52 | 0 | 0
Not completed — Subject Withdrew Consent | 0 | 47 | 0 | 0
Not completed — Non-Compliance With Study Drug | 0 | 9 | 0 | 0
Not completed — Lack of Efficacy | 0 | 136 | 0 | 0
Not completed — Pregnancy | 0 | 1 | 0 | 0
Not completed — Protocol Deviation | 0 | 9 | 0 | 0
Not completed — Physician Decision | 0 | 6 | 0 | 0
Not completed — Due to COVID-19 Restriction | 0 | 1 | 0 | 0
Not completed — Reason not Specified (not due to COVID-19 Restriction) | 0 | 11 | 0 | 0
Period: Phase C:Randomized Withdrawal (26 Weeks)
Arm/Group | Phase A: Brexpiprazole + ADT | Phase B: Brexpiprazole + ADT | Phase C: Brexpiprazole + ADT | Phase C: Placebo + ADT
Started | 0 | 0 | 240 | 249
Phase C Safety Sample (The Phase C Safety Sample included all participants who were randomized to double-blind treatment and received at least 1 dose of double-blind trial medication in Phase C.) | 0 | 0 | 240 | 248
Completed | 0 | 0 | 120 | 131
Not Completed | 0 | 0 | 120 | 118
Not completed — Lost to Follow-up | 0 | 0 | 16 | 4
Not completed — Adverse Event | 0 | 0 | 6 | 6
Not completed — Subject Withdrew Consent | 0 | 0 | 6 | 19
Not completed — Non-Compliance With Study Drug | 0 | 0 | 1 | 2
Not completed — Non-compliant Participants | 0 | 0 | 32 | 28
Not completed — Pregnancy | 0 | 0 | 1 | 0
Not completed — Lack of Efficacy (Phase C MDD Relapse) | 0 | 0 | 54 | 52
Not completed — Physician Decision | 0 | 0 | 0 | 1
Not completed — Reason not Specified (not due to COVID-19 Restriction) | 0 | 0 | 4 | 6

BASELINE CHARACTERISTICS:
Population: Enrolled Sample included all participants who signed the informed consent form and entered Phase A.
Groups:
- Phase A: Brexpiprazole + ADT: Participants received brexpiprazole 2 or 3 mg/day along with protocol-specified ADT, orally, for 6 to 8 weeks during Phase A. Participants were initially titrated to a target dose of brexpiprazole 2 mg over a 2 to 4-week period. Thereafter, participants who had not met response criteria as defined in the blinded addendum, did not have potentially dose-related AEs, and had not achieved the maximum dose of medication had their dose increased up to 3 mg.
Arm/Group | Phase A: Brexpiprazole + ADT
Number analyzed (Participants) | 1149
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.3 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 734
  Male | 415
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 110
  Not Hispanic or Latino | 968
  Unknown or Not Reported | 71
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5
  Asian | 22
  Native Hawaiian or Other Pacific Islander | 5
  Black or African American | 159
  White | 868
  More than one race | 0
  Unknown or Not Reported | 90

OUTCOME MEASURES:

1. Primary Outcome: Phase C: Time-to-Relapse by Any Criteria as Defined in Blinded Addendum
Description: Relapse criteria included:At same visit, increase in Montgomery Asberg Depression Rating Scale[MADRS] total score(10 items, 0=no symptoms to 6=severe symptoms,total score=0 to 60)of 50% from randomization and Clinical Global Impression-Severity of Illness [CGI-](8-point scale of 0=not assessed to 7=most extremely ill)score ≥4,hospitalization for depression, discontinuation for lack of efficacy/worsening of depression, active suicidality(score of ≥4 on MADRS item10 of suicidality)or yes answered on question 4 or 5 of Columbia-Suicide Severity Rating Scale[C-SSRS](Suicidal Ideation [SI] has 5 questions: wish to be dead,non-specific active suicidal thoughts,active SI with any methods [not plan]without intent to act,active SI with some intent to act without specific plan,active SI with specific plan,intent)or yes answered to any question in suicidal behavior section (5 questions:preparatory acts/behavior,aborted attempt,interrupted attempt,actual attempt[non-fatal],completed suicide).
Time Frame: Up to 14 days post last dose in Phase C (up to 28 weeks)
Population: Phase C Efficacy Sample included all participants randomized to the double-blind treatment who had taken at least one dose of investigational medicinal product (IMP) in Phase C. Overall number of participants analyzed for median time to relapse is the number of participants with impending relapse.
Measure: Median (Full Range); unit: days
Arm/Group | Phase C: Brexpiprazole + ADT | Phase C: Placebo + ADT
Number analyzed (Participants) | 54 | 51
days | 63.0 [8 to 185] | 63.0 [8 to 190]
Statistical Analysis 1: Comparison: Phase C: Brexpiprazole + ADT vs Phase C: Placebo + ADT; Test type: Superiority; p = 0.5100, Log Rank; Hazard Ratio (HR) = 1.138, 95% CI 2-sided [0.776 to 1.669] — The hazard ratio and 95% confidence interval (CI) were derived from the Cox proportional hazard model with treatment as fixed effect

2. Secondary Outcome: Phase C: Change From Baseline for Randomization Phase in Sheehan Disability Scale (SDS) Mean Total Score at Week 46
Description: The SDS is a self-rated instrument used to measure the effect of the participant's symptoms on work/school, social life, and family/home responsibilities. For each of the three items, scores range from 0 through 10. The number most representative of how much each area was disrupted by symptoms is marked along the line from 0=not at all, to 10=extremely. The SDS total score is the mean of the 3 item responses. The SDS total score ranges from 0 to 10, with higher scores indicating greater functional impairment. Baseline was defined as the last available assessment value between Week 14 and Week 20 in Phase B for this outcome measure. Analysis of covariance (ANCOVA) model was used for analysis.
Time Frame: Baseline and Week 46
Population: Phase C Efficacy Sample included all participants randomized to the double-blind treatment who had taken at least one dose of IMP in Phase C. Overall number of participants analyzed is the number of participants with data available for analyses.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Phase C: Brexpiprazole + ADT | Phase C: Placebo + ADT
Number analyzed (Participants) | 239 | 242
score on a scale | 0.72 (0.18) | 0.48 (0.18)
Statistical Analysis 1: Comparison: Phase C: Brexpiprazole + ADT vs Phase C: Placebo + ADT; Test type: Superiority; p = 0.2393, ANCOVA — P-value was derived from an ANCOVA model with treatment, pooled center as factor and Baseline value as covariance; Least Squares (LS) Mean Difference = 0.23, 95% CI 2-sided [-0.16 to 0.62]

3. Secondary Outcome: Phase C: Time-to-functional Relapse Based on SDS Criteria
Description: Time-to-functional relapse was based on a 30% increase in the SDS mean total score from Phase C Baseline, at least one SDS sub-score at 4 or greater, and an SDS total score ≥7 when all 3 sub-scores were available. The SDS is a self-rated instrument used to measure the effect of the participant's symptoms on work/school, social life, and family/home responsibilities. For each of the three items, scores range from 0 through 10. The number most representative of how much each area was disrupted by symptoms is marked along the line from 0=not at all, to 10=extremely. Higher scores of 5 and above are associated with significant functional impairment.
Time Frame: Up to 14 days post last dose in Phase C (up to 28 weeks)
Population: Phase C Efficacy Sample included all participants randomized to the double-blind treatment who had taken at least one dose of IMP in Phase C. Overall number of participants analyzed for median time to functional relapse is the number of participants with impending functional relapse.
Measure: Median (Full Range); unit: days
Arm/Group | Phase C: Brexpiprazole + ADT | Phase C: Placebo + ADT
Number analyzed (Participants) | 81 | 73
days | 36.0 [6 to 185] | 35.0 [8 to 176]
Statistical Analysis 1: Comparison: Phase C: Brexpiprazole + ADT vs Phase C: Placebo + ADT; Test type: Superiority; p = 0.3086, Log Rank; Hazard Ratio (HR) = 1.177, 95% CI 2-sided [0.857 to 1.615] — The hazard ratio and 95% CI were derived from the Cox proportional hazard model with treatment as fixed effect

4. Secondary Outcome: Phase C: Percentage of Participants Meeting Any Relapse Criteria
Description: Relapse criteria included: At the same visit, increase in MADRS total score (10 items,7-point scale of 0=no symptoms to 6=severe symptoms, total score of 0 to 60) of 50% from randomization and CGI-S (8-point scale ranging from 0=not assessed to 7=most extremely ill) score ≥4, hospitalization for depression, discontinuation for lack of efficacy/worsening of depression, active suicidality (score of ≥4 on MADRS item 10 of suicidality) or answer of yes on question 4 or 5 of C-SSRS (SI has 5 questions: wish to be dead, non-specific active suicidal thoughts, active SI with any methods [not plan] without intent to act, active SI with some intent to act without specific plan, active SI with specific plan, intent) or answer of yes to any question in suicidal behavior section (5 questions: preparatory acts/behavior, aborted attempt, interrupted attempt, actual attempt [non-fatal], completed suicide). Percentage of participants were rounded off to single decimal point.
Time Frame: Up to 26 weeks in Phase C
Population: Phase C Efficacy Sample included all participants randomized to the double-blind treatment who had taken at least one dose of IMP in Phase C.
Measure: Number; unit: percentage of participants
Arm/Group | Phase C: Brexpiprazole + ADT | Phase C: Placebo + ADT
Number analyzed (Participants) | 240 | 248
percentage of participants | 22.5 | 20.6
Statistical Analysis 1: Comparison: Phase C: Brexpiprazole + ADT vs Phase C: Placebo + ADT; Test type: Superiority; p = 0.6030, Chi-squared

5. Secondary Outcome: Phase C: Percentage of Participants Maintaining Remission
Description: Participants maintaining remission was defined as MADRS total score ≤10. The MADRS is a clinician-rated scale to assess depressive symptomatology during the preceding week. Participants were rated on 10 items (feelings of sadness, lassitude, pessimism, inner tension, suicidality, reduced sleep or appetite, difficulty concentrating, and a lack of interest) each on a 7-point scale from 0 (no symptoms) to 6 (symptoms of maximum severity). The total score ranges from 0 to 60 with a higher score indicating more depression.
Time Frame: Weeks 21, 23, 25, 29, 33, 37, 41, 45, and 46
Population: Phase C Efficacy Sample included all participants randomized to the double-blind treatment who had taken at least one dose of IMP in Phase C. Overall number of participants analyzed is the number of participants with data available for analyses. Number analyzed is the number of participants with data available for analysis at the specified timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Phase C: Brexpiprazole + ADT | Phase C: Placebo + ADT
Number analyzed (Participants) | 238 | 242
percentage of participants
  Week 21 | 90.34 | 91.3
  Week 23: number analyzed (Participants) | 230 | 237
  Week 23 | 85.22 | 82.7
  Week 25: number analyzed (Participants) | 217 | 224
  Week 25 | 84.79 | 82.6
  Week 29: number analyzed (Participants) | 189 | 200
  Week 29 | 79.89 | 85.5
  Week 33: number analyzed (Participants) | 166 | 181
  Week 33 | 88.55 | 88.4
  Week 37: number analyzed (Participants) | 149 | 164
  Week 37 | 87.92 | 89.0
  Week 41: number analyzed (Participants) | 138 | 151
  Week 41 | 84.78 | 89.4
  Week 45: number analyzed (Participants) | 118 | 127
  Week 45 | 88.14 | 89.0
  Week 46: number analyzed (Participants) | 121 | 132
  Week 46 | 90.91 | 91.7
Statistical Analysis 1: Comparison: Phase C: Brexpiprazole + ADT vs Phase C: Placebo + ADT; Week 21; Test type: Superiority; p = 0.7081, Chi-squared
Statistical Analysis 2: Comparison: Phase C: Brexpiprazole + ADT vs Phase C: Placebo + ADT; Week 23; Test type: Superiority; p = 0.4589, Chi-squared
Statistical Analysis 3: Comparison: Phase C: Brexpiprazole + ADT vs Phase C: Placebo + ADT; Week 25; Test type: Superiority; p = 0.5314, Chi-squared
Statistical Analysis 4: Comparison: Phase C: Brexpiprazole + ADT vs Phase C: Placebo + ADT; Week 29; Test type: Superiority; p = 0.1433, Chi-squared
Statistical Analysis 5: Comparison: Phase C: Brexpiprazole + ADT vs Phase C: Placebo + ADT; Week 33; Test type: Superiority; p = 0.9636, Chi-squared
Statistical Analysis 6: Comparison: Phase C: Brexpiprazole + ADT vs Phase C: Placebo + ADT; Week 37; Test type: Superiority; p = 0.7596, Chi-squared
Statistical Analysis 7: Comparison: Phase C: Brexpiprazole + ADT vs Phase C: Placebo + ADT; Week 41; Test type: Superiority; p = 0.2402, Chi-squared
Statistical Analysis 8: Comparison: Phase C: Brexpiprazole + ADT vs Phase C: Placebo + ADT; Week 45; Test type: Superiority; p = 0.8363, Chi-squared
Statistical Analysis 9: Comparison: Phase C: Brexpiprazole + ADT vs Phase C: Placebo + ADT; Week 46; Test type: Superiority; p = 0.8308, Chi-squared

6. Secondary Outcome: Phase C: Change From Baseline for Randomization Phase in MADRS Total Score at Week 46
Description: The MADRS is a clinician-rated scale to assess depressive symptomatology during the preceding week. Participants were rated on 10 items (feelings of sadness, lassitude, pessimism, inner tension, suicidality, reduced sleep or appetite, difficulty concentrating, and a lack of interest) each on a 7-point scale from 0 (no symptoms) to 6 (symptoms of maximum severity). The total score ranges from 0 to 60 with a higher score indicating more depression. A positive change from Baseline indicates worsening of symptoms. Baseline was defined as the last available assessment value in Phase B for this outcome measure. ANCOVA model was used for analysis.
Time Frame: Baseline and Week 46
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Phase C: Brexpiprazole + ADT | Phase C: Placebo + ADT
Number analyzed (Participants) | 240 | 247
score on a scale | 4.09 (0.75) | 4.21 (0.73)
Statistical Analysis 1: Comparison: Phase C: Brexpiprazole + ADT vs Phase C: Placebo + ADT; Test type: Superiority; p = 0.8806, ANCOVA; P-value was derived from an ANCOVA model with treatment, pooled center as factor and Baseline value as covariance; LS Mean Difference = -0.12, 95% CI 2-sided [-1.73 to 1.49]

7. Secondary Outcome: Phase C: Change From Baseline for Randomization Phase in CGI-S Score at Week 46
Description: The CGI -S was used to rate the severity of illness for each participant on an 8-point scale ranging from 0 to 7 where 0=not assessed, 1=normal, not at all ill, 2=borderline mentally ill, 3=mildly ill, 4=moderately ill, 5=markedly ill, 6=severely ill, and 7=among the most extremely ill participants. A positive change from Baseline indicates worsening of illness. Baseline was defined as the last available assessment value in Phase B for this outcome measure. ANCOVA model was used for analysis.
Time Frame: Baseline and Week 46
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Phase C: Brexpiprazole + ADT | Phase C: Placebo + ADT
Number analyzed (Participants) | 240 | 247
score on a scale | 0.56 (0.10) | 0.53 (0.09)
Statistical Analysis 1: Comparison: Phase C: Brexpiprazole + ADT vs Phase C: Placebo + ADT; Test type: Superiority; p = 0.7956, ANCOVA; P-value was derived from an ANCOVA model with treatment, pooled center as factor and Baseline value as covariance; LS Mean Difference = 0.03, 95% CI 2-sided [-0.18 to 0.24]

8. Secondary Outcome: Phase C: Change From Baseline for Randomization Phase in Each of the SDS Individual Item Scores at Week 46
Description: The SDS is a self-rated instrument used to measure the effect of the participant's symptoms on work/school, social life, and family/home responsibilities. For each of the three items, scores range from 0 through 10. The number most representative of how much each area was disrupted by symptoms is marked along the line from 0=not at all, to 10=extremely. Higher scores of 5 and above are associated with significant functional impairment. A positive change from Baseline indicates worsening of symptoms impacting each area. Baseline was defined as the last available assessment value between Week 14 and Week 20 in Phase B for this outcome measure. ANCOVA model was used for analysis.
Time Frame: Baseline and Week 46
Population: Phase C Efficacy Sample included all participants randomized to the double-blind treatment who had taken at least one dose of IMP in Phase C. Overall number of participants analyzed is the number of participants with data available for analyses. Number analyzed is the number of participants with data available for analysis for the specified category.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Phase C: Brexpiprazole + ADT | Phase C: Placebo + ADT
Number analyzed (Participants) | 239 | 244
score on a scale
  Work/School: number analyzed (Participants) | 195 | 197
  Work/School | 0.46 (0.22) | 0.31 (0.23)
  Social Life | 0.91 (0.19) | 0.56 (0.19)
  Family Life: number analyzed (Participants) | 239 | 242
  Family Life | 0.78 (0.19) | 0.52 (0.19)
Statistical Analysis 1: Comparison: Phase C: Brexpiprazole + ADT vs Phase C: Placebo + ADT; SDS Individual Item: Work/School; Test type: Superiority; p = 0.5223, ANCOVA — P-value was derived from an ANCOVA model with treatment, pooled center as factor and Baseline value as covariance; LS Mean Difference = 0.15, 95% CI 2-sided [-0.31 to 0.61]
Statistical Analysis 2: Comparison: Phase C: Brexpiprazole + ADT vs Phase C: Placebo + ADT; SDS Individual Item: Social Life; Test type: Superiority; p = 0.0904, ANCOVA — P-value was derived from an ANCOVA model with treatment, pooled center as factor and Baseline value as covariance; LS Mean Difference = 0.36, 95% CI 2-sided [-0.06 to 0.77]
Statistical Analysis 3: Comparison: Phase C: Brexpiprazole + ADT vs Phase C: Placebo + ADT; SDS Individual Item: Family Life; Test type: Superiority; p = 0.2289, ANCOVA — P-value was derived from an ANCOVA model with treatment, pooled center as factor and Baseline value as covariance; LS Mean Difference = 0.25, 95% CI 2-sided [-0.16 to 0.67]

ADVERSE EVENTS:
Time Frame: From first dose of study drug to 21 days after the last dose (Up to 49 weeks)
Description: All-cause Mortality: Enrolled Sample included all participants who signed informed consent form and entered Phase A.
  Serious and Other AEs: Phase A Safety Sample=all participants who received at least 1 dose of brexpiprazole in Phase A. Phase B Safety Sample=all participants who received at least 1 dose of brexpiprazole in Phase B. Phase C Safety Sample=all participants who were randomized to double-blind treatment and received at least one dose of double-blind trial medication in Phase C.
Arm/Group | Phase A: Brexpiprazole + ADT | Phase B: Brexpiprazole + ADT | Phase C: Brexpiprazole + ADT | Phase C: Placebo + ADT
All-Cause Mortality (participants affected / at risk) | 1/1149 | 0/766 | 0/240 | 0/249
Serious Adverse Events (participants affected / at risk) | 10/1136 | 12/765 | 1/240 | 3/248
Other Adverse Events (participants affected / at risk) | 398/1136 | 163/765 | 25/240 | 13/248
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase A: Brexpiprazole + ADT (N=1136) | Phase B: Brexpiprazole + ADT (N=765) | Phase C: Brexpiprazole + ADT (N=240) | Phase C: Placebo + ADT (N=248)
Cataract (Eye disorders) | 0 | 0 | 0 | 1
Anaphylactic shock (Immune system disorders) | 0 | 0 | 1 | 0
Dislocation of vertebra (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Epicondylitis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Acute hepatic failure (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 1 | 0 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Akathisia (Nervous system disorders) | 1 | 0 | 0 | 0
Cervicobrachial syndrome (Nervous system disorders) | 1 | 0 | 0 | 0
Major depression (Psychiatric disorders) | 1 | 0 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase A: Brexpiprazole + ADT (N=1136) | Phase B: Brexpiprazole + ADT (N=765) | Phase C: Brexpiprazole + ADT (N=240) | Phase C: Placebo + ADT (N=248)
Weight increased (Investigations) | 0 | 122 | 25 | 13
Headache (Nervous system disorders) | 113 | 41 | 0 | 0
Nausea (Gastrointestinal disorders) | 64 | 0 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 60 | 0 | 0 | 0
Akathisia (Nervous system disorders) | 109 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 90 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 72 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-07-16): https://cdn.clinicaltrials.gov/large-docs/91/NCT03538691/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-13): https://cdn.clinicaltrials.gov/large-docs/91/NCT03538691/SAP_001.pdf